CLINICAL TRIAL: NCT04558125
Title: Low-Dose Tenecteplase in Covid-19 Patients With Acute Pulmonary Embolism: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Low-Dose Tenecteplase in Covid-19 Diagnosed With Pulmonary Embolism
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Identification of eligible patients was slower than anticipated.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Victor Tapson, MD, Professor of Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ML42522
Record Dates: First submitted 2020-09-19; First posted 2020-09-22 (Actual); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Embolism; COVID
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tenecteplase; Enoxaparin; Heparin, Low-Molecular-Weight; enoxaparin sodium; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low-dose TNKase and Standard of Care Anticoagulation (Experimental): 1. TNKase (0.25 mg/kg) bolus Other names: Tenecteplase, TNK
  2. Standard of care anticoagulation (heparin or enoxaparin)
  Interventions: Drug: TNKase; Drug: Enoxaparin
- Placebo and and Standard of Care Anticoagulation (Active Comparator): 1. Placebo bolus (intravenous syringe identical to that of TNK )
  2. Standard of care anticoagulation (heparin or enoxaparin)
  Interventions: Drug: Placebo; Drug: Enoxaparin

INTERVENTIONS:
Drug: TNKase — Tenecteplase (0.25 mg/kg) supplied by Genentech, Inc. as a sterile, lyophilized powder, diluted with 10mL sterile water.
  Other Names: Tenecteplase; TNK
  Arms: Low-dose TNKase and Standard of Care Anticoagulation
Drug: Placebo — Placebo to match supplied by Genentech, Inc. as a sterile, lyophilized powder, diluted with 10mL sterile water.
  Arms: Placebo and and Standard of Care Anticoagulation
Drug: Enoxaparin — All participants must also receive standard of care anticoagulation therapy.
  Other Names: Low molecular weight heparin; Lovenox; Enoxaparin sodium; Heparin; Heparin sodium

SUMMARY:
* There is a knowledge gap associated with the management of patients with COVID-19 lung injury and a laboratory picture compatible with disseminated intravascular coagulation (DIC). Clinical data to date support that COVID-19 is associated with a prothrombotic state that is not simply explained by an influx of more critically ill individuals.
* These patients suffer from severe respiratory failure; hypoxemia and ventilator dependence are the primary concerns; ARDS with respiratory failure is frequently the cause of death. Macroscopic and probable microvascular thromboembolic events are a major concern in this population.
* When DIC is associated with COVID-19, it predicts a very poor prognosis.
* This study will evaluate the clinical efficacy and safety of low-dose IV bolus tenecteplase (TNK) together with anticoagulation compared with control patients on therapeutic anticoagulation alone in hospitalized adults diagnosed with COVID-19 and acute intermediate-risk PE.
* Prospective, multicenter, randomized two-arm trial enrolling consecutive patients who meet enrollment criteria.
* The study will generate evidence that low-dose TNK together with anticoagulation is beneficial in these patients

DETAILED DESCRIPTION:
This is a prospective, double-blind, placebo-controlled study randomizing patients with acute intermediate-risk PE who meet enrollment criteria in a 2:1 manner into intervention (TNK) versus placebo arms, respectively. There will be up to 6 sites. After 18 patients are enrolled, a safety assessment will be performed by an independent Data and Safety Monitoring Board, and if a safety issue arises, it will be considered and discussed among the investigators. The planned sample size is 45 patients (30 treatment and 15 control). Subjects will be assessed daily while hospitalized. Subjects discharged from the hospital will be asked to attend study visits at Days 14 and 30 (telephone / telemedicine, clinic or inpatient ward).

The overall objective of the study is to evaluate the clinical efficacy and safety of IV bolus tenecteplase (TNK) and therapeutic anticoagulation compared with placebo and therapeutic anticoagulation in hospitalized adults diagnosed with COVID-19 infection and acute intermediate-risk PE.

Written informed consent for participation in the study must be obtained before performing any study-related procedures (including screening evaluations). Informed Consent Forms for enrolled patients and for patients who are not subsequently enrolled will be maintained at the study site.

After informed consent is obtained, screening assessment will be completed to confirm a patient's eligibility for participation in the study. The screening visit will include medical history, physical exam and vital signs. Standard of care (SOC). labs will be reviewed. These may include INR, aPTT, PT (if patient is currently taking an anticoagulant), CBC with diff, comprehensive chemistry panel, D-dimer and Ferritin. The results of the SARS-CoV-2 will be documented. If subject is in child-bearing age and a pregnancy test was not done for SOC, a urine pregnancy test will be performed. Electrocadiogram and CTA will be reviewed.

If the patient is determined to be eligible, the study site will obtain the patient's medical record number/unique patient identification number, and treatment assignment to either interventional (TNK) or placebo will be randomly determined. Patients will be allocated to the interventional versus placebo arms in a 2:1 manner as per a computer-generated randomization schedule using permuted blocks of random sizes. The block sizes will not be disclosed to ensure concealment. A total of 30 TNK subjects versus 15 placebo controls will be enrolled.

Before the study drug/placebo is administered, the following labs will be drawn CBC with diff, comprehensive metabolic panel, CRP, Ferritin, IL-6, Fibrinogen, D-dimer, PT/PTT, LDH, lactate, troponin, creatinine kinase, and Thromboelastography (TEG). Vital signs and echocardiogram will be obtained. Shock Index will be calculated, then the infusion will begin.

Within 10 minutes (+ 5min) of infusion, a second TEG will be collected. At 6 hours after the infusion, a second Shock Index will be calculated. At 24+/- 6 hours after the bolus, a physical exam will be performed, vital signs will be collected, an echocardiogram will be performed and D-dimer, CRP, IL-6, and Ferritin will be done. TEG will be an optional addition to the 24-hour labs. Daily safety labs will include CBC and chemistry panel. SOC lab results will be collected from the chart.

Patients will have follow-up visits on Day 14 +/- 2 days and Day 30 +/- 4 days. These visits may take place via televisit or in person. Data will be collected on adverse events, vital signs and new concomitant medications. Safety labs will be obtained if visit occurs in person.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female adult ≥18 years of age, but < 75 years of age at time of enrollment.
2. Laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen < 28 days prior to randomization, OR person under investigation (PUI) of COVID-19 with pulmonary infiltrates and elevated ferritin and CRP level.
3. Acute intermediate-risk pulmonary embolism defined as:

   * Presence of acute pulmonary embolism confirmed by diagnostic imaging (computed tomographic angiography, ventilation-perfusion scan, or invasive pulmonary angiography) AND
   * Presence of clot burden with at least one lobar artery involved OR bilateral with at least segmental branches OR unilateral clot in at least multiple segmental branches.
4. Subject (or legally authorized representative) provides written informed consent prior to the performance of any study procedures.
5. In the Investigator's judgement, patient has the ability to comply with the study protocol, and understands and agrees to comply with planned TNK bolus versus placebo.

Exclusion Criteria:

1. Anticipated transfer to another hospital (which is not a study site) within 72 hours
2. Allergy or contraindications to TNK
3. Contraindications to systemic anticoagulation
4. Active bleeding
5. Known significant bleeding risk (although recent exposure to aspirin or any other antiplatelet therapy is not an exclusion criterion). While there is no specific hemoglobin cut-off value for enrollment, Investigators will gauge the severity / stability of the Hgb and exclude patients deemed inappropriate.
6. Major GI or GU bleed within the past 3 weeks
7. History of hemorrhagic stroke
8. History of acute ischemic stroke in the last 90 days
9. High-risk (massive) acute PE (PE associated with hypotension (systolic BP < 90 mmHg for > 15 min).
10. PE associated with syncope and any degree of head trauma
11. PE meeting criteria for intermediate-risk PE and thus for enrollment, but with clinical evidence of deterioration such that the Investigator deems the patient not appropriate for enrollment.
12. Administration of thrombolytic agent within the previous 7 days
13. Pulmonary thrombectomy within the previous 30 days
14. Uncontrolled hypertension defined as systolic blood pressure >180 mm Hg and/or diastolic blood pressure >110 mm Hg at randomization
15. Severe ARDS (P/F ratio < 100)
16. Platelet count lower than 80,000/mm3
17. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; recent oral anticoagulant therapy with INR >1.7
18. Arterial puncture at a non-compressible site within the past 5 days
19. Prior brain surgery
20. Severe trauma in the prior 2 weeks
21. Major surgery in the prior 2 weeks
22. Brain malignancy / metastases, brain tumor in past 5 years
23. Brain AVM or ruptured aneurysm at any time
24. Acute myocardial infarction or history of myocardial infarction within the past 3 weeks or cardiac arrest during hospitalization
25. Cardiac tamponade
26. Lumbar puncture with in past 7 days
27. Known abdominal or thoracic aneurysm
28. Acute or chronic renal failure requiring dialysis
29. Chronic liver failure (acutely elevated liver function tests not an exclusion criterion)
30. Bacterial endocarditis at time of study entry
31. Seizure during pre-hospital course or during hospitalization for COVID-19
32. Currently on ECMO
33. Pregnancy, lactation or parturition within the previous 30 days
34. Patients, in whom, in the opinion of the Investigator, are critically ill from concomitant comorbid cardiopulmonary disease, and unlikely to benefit.
35. Any other condition that the Investigator felt would place the patient at increased risk if the investigational therapy were initiated
36. Previous enrollment in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor E Tapson, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morens DM, Daszak P, Taubenberger JK. Escaping Pandora's Box - Another Novel Coronavirus. N Engl J Med. 2020 Apr 2;382(14):1293-1295. doi: 10.1056/NEJMp2002106. Epub 2020 Feb 26. No abstract available. PMID 32101660
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Han H, Yang L, Liu R, Liu F, Wu KL, Li J, Liu XH, Zhu CL. Prominent changes in blood coagulation of patients with SARS-CoV-2 infection. Clin Chem Lab Med. 2020 Jun 25;58(7):1116-1120. doi: 10.1515/cclm-2020-0188. PMID 32172226
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Sebag SC, Bastarache JA, Ware LB. Therapeutic modulation of coagulation and fibrinolysis in acute lung injury and the acute respiratory distress syndrome. Curr Pharm Biotechnol. 2011 Sep;12(9):1481-96. doi: 10.2174/138920111798281171. PMID 21401517
- [Background] Ware LB, Bastarache JA, Wang L. Coagulation and fibrinolysis in human acute lung injury--new therapeutic targets? Keio J Med. 2005 Sep;54(3):142-9. doi: 10.2302/kjm.54.142. PMID 16237276
- [Background] Finigan JH. The coagulation system and pulmonary endothelial function in acute lung injury. Microvasc Res. 2009 Jan;77(1):35-8. doi: 10.1016/j.mvr.2008.09.002. Epub 2008 Sep 18. PMID 18938186
- [Background] Idell S, Koenig KB, Fair DS, Martin TR, McLarty J, Maunder RJ. Serial abnormalities of fibrin turnover in evolving adult respiratory distress syndrome. Am J Physiol. 1991 Oct;261(4 Pt 1):L240-8. doi: 10.1152/ajplung.1991.261.4.L240. PMID 1928357
- [Background] Prabhakaran P, Ware LB, White KE, Cross MT, Matthay MA, Olman MA. Elevated levels of plasminogen activator inhibitor-1 in pulmonary edema fluid are associated with mortality in acute lung injury. Am J Physiol Lung Cell Mol Physiol. 2003 Jul;285(1):L20-8. doi: 10.1152/ajplung.00312.2002. Epub 2003 May 2. PMID 12730079
- [Background] Ware LB, Matthay MA, Parsons PE, Thompson BT, Januzzi JL, Eisner MD; National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome Clinical Trials Network. Pathogenetic and prognostic significance of altered coagulation and fibrinolysis in acute lung injury/acute respiratory distress syndrome. Crit Care Med. 2007 Aug;35(8):1821-8. doi: 10.1097/01.CCM.0000221922.08878.49. PMID 17667242
- [Background] Moalli R, Doyle JM, Tahhan HR, Hasan FM, Braman SS, Saldeen T. Fibrinolysis in critically ill patients. Am Rev Respir Dis. 1989 Aug;140(2):287-93. doi: 10.1164/ajrccm/140.2.287. PMID 2504087
- [Background] Texereau J, Pene F, Chiche JD, Rousseau C, Mira JP. Importance of hemostatic gene polymorphisms for susceptibility to and outcome of severe sepsis. Crit Care Med. 2004 May;32(5 Suppl):S313-9. doi: 10.1097/01.ccm.0000126363.46191.dc. PMID 15118537
- [Background] Hardaway RM, Williams CH, Marvasti M, Farias M, Tseng A, Pinon I, Yanez D, Martinez M, Navar J. Prevention of adult respiratory distress syndrome with plasminogen activator in pigs. Crit Care Med. 1990 Dec;18(12):1413-8. doi: 10.1097/00003246-199012000-00021. PMID 2123144
- [Background] Hart DA, Whidden P, Green F, Henkin J, Woods DE. Partial reversal of established bleomycin-induced pulmonary fibrosis by rh-urokinase in a rat model. Clin Invest Med. 1994 Apr;17(2):69-76. PMID 7516275
- [Background] Hardaway RM, Harke H, Tyroch AH, Williams CH, Vazquez Y, Krause GF. Treatment of severe acute respiratory distress syndrome: a final report on a phase I study. Am Surg. 2001 Apr;67(4):377-82. PMID 11308009
- [Background] Stringer KA, Hybertson BM, Cho OJ, Cohen Z, Repine JE. Tissue plasminogen activator (tPA) inhibits interleukin-1 induced acute lung leak. Free Radic Biol Med. 1998 Jul 15;25(2):184-8. doi: 10.1016/s0891-5849(98)00047-1. PMID 9667494
- [Background] Burgos AM, Saver JL. Evidence that Tenecteplase Is Noninferior to Alteplase for Acute Ischemic Stroke: Meta-Analysis of 5 Randomized Trials. Stroke. 2019 Aug;50(8):2156-2162. doi: 10.1161/STROKEAHA.119.025080. Epub 2019 Jul 18. PMID 31318627
- [Background] Guillermin A, Yan DJ, Perrier A, Marti C. Safety and efficacy of tenecteplase versus alteplase in acute coronary syndrome: a systematic review and meta-analysis of randomized trials. Arch Med Sci. 2016 Dec 1;12(6):1181-1187. doi: 10.5114/aoms.2016.58929. Epub 2016 Mar 31. PMID 27904506
- [Background] Meyer G, Vicaut E, Danays T, Agnelli G, Becattini C, Beyer-Westendorf J, Bluhmki E, Bouvaist H, Brenner B, Couturaud F, Dellas C, Empen K, Franca A, Galie N, Geibel A, Goldhaber SZ, Jimenez D, Kozak M, Kupatt C, Kucher N, Lang IM, Lankeit M, Meneveau N, Pacouret G, Palazzini M, Petris A, Pruszczyk P, Rugolotto M, Salvi A, Schellong S, Sebbane M, Sobkowicz B, Stefanovic BS, Thiele H, Torbicki A, Verschuren F, Konstantinides SV; PEITHO Investigators. Fibrinolysis for patients with intermediate-risk pulmonary embolism. N Engl J Med. 2014 Apr 10;370(15):1402-11. doi: 10.1056/NEJMoa1302097. PMID 24716681
- [Background] Becattini C, Agnelli G, Salvi A, Grifoni S, Pancaldi LG, Enea I, Balsemin F, Campanini M, Ghirarduzzi A, Casazza F; TIPES Study Group. Bolus tenecteplase for right ventricle dysfunction in hemodynamically stable patients with pulmonary embolism. Thromb Res. 2010 Mar;125(3):e82-6. doi: 10.1016/j.thromres.2009.09.017. Epub 2009 Oct 14. PMID 19833379
- [Background] Caldicott D, Parasivam S, Harding J, Edwards N, Bochner F. Tenecteplase for massive pulmonary embolus. Resuscitation. 2002 Nov;55(2):211-3. doi: 10.1016/s0300-9572(02)00171-5. PMID 12413760
- [Background] Burkart DJ, Borsa JJ, Anthony JP, Thurlo SR. Thrombolysis of occluded peripheral arteries and veins with tenecteplase: a pilot study. J Vasc Interv Radiol. 2002 Nov;13(11):1099-102. doi: 10.1016/s1051-0443(07)61950-2. PMID 12427808
- [Background] Thachil J, Tang N, Gando S, Falanga A, Cattaneo M, Levi M, Clark C, Iba T. ISTH interim guidance on recognition and management of coagulopathy in COVID-19. J Thromb Haemost. 2020 May;18(5):1023-1026. doi: 10.1111/jth.14810. Epub 2020 Apr 27. No abstract available. PMID 32338827
- [Background] Tang N, Bai H, Chen X, Gong J, Li D, Sun Z. Anticoagulant treatment is associated with decreased mortality in severe coronavirus disease 2019 patients with coagulopathy. J Thromb Haemost. 2020 May;18(5):1094-1099. doi: 10.1111/jth.14817. Epub 2020 Apr 27. PMID 32220112
- [Background] Paranjpe I, Fuster V, Lala A, Russak AJ, Glicksberg BS, Levin MA, Charney AW, Narula J, Fayad ZA, Bagiella E, Zhao S, Nadkarni GN. Association of Treatment Dose Anticoagulation With In-Hospital Survival Among Hospitalized Patients With COVID-19. J Am Coll Cardiol. 2020 Jul 7;76(1):122-124. doi: 10.1016/j.jacc.2020.05.001. Epub 2020 May 6. No abstract available. PMID 32387623
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Background] Poissy J, Goutay J, Caplan M, Parmentier E, Duburcq T, Lassalle F, Jeanpierre E, Rauch A, Labreuche J, Susen S; Lille ICU Haemostasis COVID-19 Group. Pulmonary Embolism in Patients With COVID-19: Awareness of an Increased Prevalence. Circulation. 2020 Jul 14;142(2):184-186. doi: 10.1161/CIRCULATIONAHA.120.047430. Epub 2020 Apr 24. No abstract available. PMID 32330083
- [Background] Wichmann D, Sperhake JP, Lutgehetmann M, Steurer S, Edler C, Heinemann A, Heinrich F, Mushumba H, Kniep I, Schroder AS, Burdelski C, de Heer G, Nierhaus A, Frings D, Pfefferle S, Becker H, Bredereke-Wiedling H, de Weerth A, Paschen HR, Sheikhzadeh-Eggers S, Stang A, Schmiedel S, Bokemeyer C, Addo MM, Aepfelbacher M, Puschel K, Kluge S. Autopsy Findings and Venous Thromboembolism in Patients With COVID-19: A Prospective Cohort Study. Ann Intern Med. 2020 Aug 18;173(4):268-277. doi: 10.7326/M20-2003. Epub 2020 May 6. PMID 32374815
- [Background] Albers GW, Marks MP, Kemp S, Christensen S, Tsai JP, Ortega-Gutierrez S, McTaggart RA, Torbey MT, Kim-Tenser M, Leslie-Mazwi T, Sarraj A, Kasner SE, Ansari SA, Yeatts SD, Hamilton S, Mlynash M, Heit JJ, Zaharchuk G, Kim S, Carrozzella J, Palesch YY, Demchuk AM, Bammer R, Lavori PW, Broderick JP, Lansberg MG; DEFUSE 3 Investigators. Thrombectomy for Stroke at 6 to 16 Hours with Selection by Perfusion Imaging. N Engl J Med. 2018 Feb 22;378(8):708-718. doi: 10.1056/NEJMoa1713973. Epub 2018 Jan 24. PMID 29364767
- [Background] Benedict CR, Refino CJ, Keyt BA, Pakala R, Paoni NF, Thomas GR, Bennett WF. New variant of human tissue plasminogen activator (TPA) with enhanced efficacy and lower incidence of bleeding compared with recombinant human TPA. Circulation. 1995 Nov 15;92(10):3032-40. doi: 10.1161/01.cir.92.10.3032. PMID 7586274
- [Background] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Background] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Background] Bivard A, Huang X, McElduff P, Levi CR, Campbell BC, Cheripelli BK, Kalladka D, Moreton FC, Ford I, Bladin CF, Davis SM, Donnan GA, Muir KW, Parsons MW. Impact of Computed Tomography Perfusion Imaging on the Response to Tenecteplase in Ischemic Stroke: Analysis of 2 Randomized Controlled Trials. Circulation. 2017 Jan 31;135(5):440-448. doi: 10.1161/CIRCULATIONAHA.116.022582. Epub 2016 Dec 13. PMID 27965285
- [Background] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Background] From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO); Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Shazam Hussain M, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke. Int J Stroke. 2018 Aug;13(6):612-632. doi: 10.1177/1747493018778713. Epub 2018 May 22. No abstract available. PMID 29786478
- [Background] Churilov L, Arnup S, Johns H, Leung T, Roberts S, Campbell BC, Davis SM, Donnan GA. An improved method for simple, assumption-free ordinal analysis of the modified Rankin Scale using generalized odds ratios. Int J Stroke. 2014 Dec;9(8):999-1005. doi: 10.1111/ijs.12364. Epub 2014 Sep 4. PMID 25196780
- [Background] Coutts SB, Dubuc V, Mandzia J, Kenney C, Demchuk AM, Smith EE, Subramaniam S, Goyal M, Patil S, Menon BK, Barber PA, Dowlatshahi D, Field T, Asdaghi N, Camden MC, Hill MD; TEMPO-1 Investigators. Tenecteplase-tissue-type plasminogen activator evaluation for minor ischemic stroke with proven occlusion. Stroke. 2015 Mar;46(3):769-74. doi: 10.1161/STROKEAHA.114.008504. Epub 2015 Feb 12. PMID 25677596
- [Background] DeMets DL, Lan KK. Interim analysis: the alpha spending function approach. Stat Med. 1994 Jul 15-30;13(13-14):1341-52; discussion 1353-6. doi: 10.1002/sim.4780131308. PMID 7973215
- [Background] Emberson J, Lees KR, Lyden P, Blackwell L, Albers G, Bluhmki E, Brott T, Cohen G, Davis S, Donnan G, Grotta J, Howard G, Kaste M, Koga M, von Kummer R, Lansberg M, Lindley RI, Murray G, Olivot JM, Parsons M, Tilley B, Toni D, Toyoda K, Wahlgren N, Wardlaw J, Whiteley W, del Zoppo GJ, Baigent C, Sandercock P, Hacke W; Stroke Thrombolysis Trialists' Collaborative Group. Effect of treatment delay, age, and stroke severity on the effects of intravenous thrombolysis with alteplase for acute ischaemic stroke: a meta-analysis of individual patient data from randomised trials. Lancet. 2014 Nov 29;384(9958):1929-35. doi: 10.1016/S0140-6736(14)60584-5. Epub 2014 Aug 5. PMID 25106063
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Background] Haley EC Jr, Lyden PD, Johnston KC, Hemmen TM; TNK in Stroke Investigators. A pilot dose-escalation safety study of tenecteplase in acute ischemic stroke. Stroke. 2005 Mar;36(3):607-12. doi: 10.1161/01.STR.0000154872.73240.e9. Epub 2005 Feb 3. PMID 15692126
- [Background] Haley EC Jr, Thompson JL, Grotta JC, Lyden PD, Hemmen TG, Brown DL, Fanale C, Libman R, Kwiatkowski TG, Llinas RH, Levine SR, Johnston KC, Buchsbaum R, Levy G, Levin B; Tenecteplase in Stroke Investigators. Phase IIB/III trial of tenecteplase in acute ischemic stroke: results of a prematurely terminated randomized clinical trial. Stroke. 2010 Apr;41(4):707-11. doi: 10.1161/STROKEAHA.109.572040. Epub 2010 Feb 25. PMID 20185783
- [Background] Howard G, Waller JL, Voeks JH, Howard VJ, Jauch EC, Lees KR, Nichols FT, Rahlfs VW, Hess DC. A simple, assumption-free, and clinically interpretable approach for analysis of modified Rankin outcomes. Stroke. 2012 Mar;43(3):664-9. doi: 10.1161/STROKEAHA.111.632935. Epub 2012 Feb 16. PMID 22343650
- [Background] Huang X, Cheripelli BK, Lloyd SM, Kalladka D, Moreton FC, Siddiqui A, Ford I, Muir KW. Alteplase versus tenecteplase for thrombolysis after ischaemic stroke (ATTEST): a phase 2, randomised, open-label, blinded endpoint study. Lancet Neurol. 2015 Apr;14(4):368-76. doi: 10.1016/S1474-4422(15)70017-7. Epub 2015 Feb 26. PMID 25726502
- [Background] Huang X, MacIsaac R, Thompson JL, Levin B, Buchsbaum R, Haley EC Jr, Levi C, Campbell B, Bladin C, Parsons M, Muir KW. Tenecteplase versus alteplase in stroke thrombolysis: An individual patient data meta-analysis of randomized controlled trials. Int J Stroke. 2016 Jul;11(5):534-43. doi: 10.1177/1747493016641112. Epub 2016 Apr 5. PMID 27048693
- [Background] Jovin TG, Liebeskind DS, Gupta R, Rymer M, Rai A, Zaidat OO, Abou-Chebl A, Baxter B, Levy EI, Barreto A, Nogueira RG. Imaging-based endovascular therapy for acute ischemic stroke due to proximal intracranial anterior circulation occlusion treated beyond 8 hours from time last seen well: retrospective multicenter analysis of 237 consecutive patients. Stroke. 2011 Aug;42(8):2206-11. doi: 10.1161/STROKEAHA.110.604223. Epub 2011 Jul 21. PMID 21778444
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Background] Kate M, Wannamaker R, Kamble H, Riaz P, Gioia LC, Buck B, Jeerakathil T, Smyth P, Shuaib A, Emery D, Butcher K. Penumbral Imaging-Based Thrombolysis with Tenecteplase Is Feasible up to 24 Hours after Symptom Onset. J Stroke. 2018 Jan;20(1):122-130. doi: 10.5853/jos.2017.00178. Epub 2018 Jan 31. PMID 29402060
- [Background] Lansberg MG, Cereda CW, Mlynash M, Mishra NK, Inoue M, Kemp S, Christensen S, Straka M, Zaharchuk G, Marks MP, Bammer R, Albers GW; Diffusion and Perfusion Imaging Evaluation for Understanding Stroke Evolution 2 (DEFUSE 2) Study Investigators. Response to endovascular reperfusion is not time-dependent in patients with salvageable tissue. Neurology. 2015 Aug 25;85(8):708-14. doi: 10.1212/WNL.0000000000001853. Epub 2015 Jul 29. PMID 26224727
- [Background] Logallo N, Kvistad CE, Thomassen L. Therapeutic Potential of Tenecteplase in the Management of Acute Ischemic Stroke. CNS Drugs. 2015;29(10):811-8. doi: 10.1007/s40263-015-0280-9. PMID 26387127
- [Background] Logallo N, Novotny V, Assmus J, Kvistad CE, Alteheld L, Ronning OM, Thommessen B, Amthor KF, Ihle-Hansen H, Kurz M, Tobro H, Kaur K, Stankiewicz M, Carlsson M, Morsund A, Idicula T, Aamodt AH, Lund C, Naess H, Waje-Andreassen U, Thomassen L. Tenecteplase versus alteplase for management of acute ischaemic stroke (NOR-TEST): a phase 3, randomised, open-label, blinded endpoint trial. Lancet Neurol. 2017 Oct;16(10):781-788. doi: 10.1016/S1474-4422(17)30253-3. Epub 2017 Aug 2. PMID 28780236
- [Background] Nogueira RG, Jadhav AP, Haussen DC, Bonafe A, Budzik RF, Bhuva P, Yavagal DR, Ribo M, Cognard C, Hanel RA, Sila CA, Hassan AE, Millan M, Levy EI, Mitchell P, Chen M, English JD, Shah QA, Silver FL, Pereira VM, Mehta BP, Baxter BW, Abraham MG, Cardona P, Veznedaroglu E, Hellinger FR, Feng L, Kirmani JF, Lopes DK, Jankowitz BT, Frankel MR, Costalat V, Vora NA, Yoo AJ, Malik AM, Furlan AJ, Rubiera M, Aghaebrahim A, Olivot JM, Tekle WG, Shields R, Graves T, Lewis RJ, Smith WS, Liebeskind DS, Saver JL, Jovin TG; DAWN Trial Investigators. Thrombectomy 6 to 24 Hours after Stroke with a Mismatch between Deficit and Infarct. N Engl J Med. 2018 Jan 4;378(1):11-21. doi: 10.1056/NEJMoa1706442. Epub 2017 Nov 11. PMID 29129157
- [Background] Parsons MW, Levi CR. Reperfusion trials for acute ischaemic stroke. Lancet. 2012 Aug 25;380(9843):706-8. doi: 10.1016/S0140-6736(12)61043-5. Epub 2012 Jun 28. No abstract available. PMID 22748819
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Background] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Devlin TG, Lopes DK, Reddy V, du Mesnil de Rochemont R, Jahan R; SWIFT PRIME Investigators. Solitaire with the Intention for Thrombectomy as Primary Endovascular Treatment for Acute Ischemic Stroke (SWIFT PRIME) trial: protocol for a randomized, controlled, multicenter study comparing the Solitaire revascularization device with IV tPA with IV tPA alone in acute ischemic stroke. Int J Stroke. 2015 Apr;10(3):439-48. doi: 10.1111/ijs.12459. PMID 25777831
- [Background] Ovbiagele B, Goldstein LB, Higashida RT, Howard VJ, Johnston SC, Khavjou OA, Lackland DT, Lichtman JH, Mohl S, Sacco RL, Saver JL, Trogdon JG; American Heart Association Advocacy Coordinating Committee and Stroke Council. Forecasting the future of stroke in the United States: a policy statement from the American Heart Association and American Stroke Association. Stroke. 2013 Aug;44(8):2361-75. doi: 10.1161/STR.0b013e31829734f2. Epub 2013 May 22. PMID 23697546
- See also: Stroke Early Management Guidelines — http://www.acc.org/latest-in-cardiology/ten-points-to-remember/2018/01/29/12/45/2018-guidelines-for-the-early-management-of-stroke
- See also: TEG max clot strength is consistently elevated and may be predictive of COVID-19 status at the time of ICU admission — https://doi.org/10.1101/2020.04.30.20076703
- See also: A randomized trial of anticoagulation strategies in COVID-19 — https://clinicaltrials.gov/ct2/show/NCT04359277
- See also: Preventing COVID-19 complications with low- and high-dose anticoagulation (COVID-HEP) — https://clinicaltrials.gov/ct2/show/NCT04345848
- See also: Trial evaluating efficacy and safety of anticoagulation in patients with COVID-19 infection, nested in the Corimmuno-19 Cohort (CORIMMUNO-COAG) — https://clinicaltrials.gov/ct2/show/NCT04344756
- See also: Risk assessment of venous thromboembolism and bleeding in COVID-19 patients — https://www.researchgate.net/publication/340140994_Risk_assessment_of_venous_thromboembolism_and_bleeding_in_COVID-19_patients
- See also: Clinical pathology of critical patient with novel coronavirus pneumonia (COVID-19) — https://www.researchgate.net/publication/339939319_Clinical_Pathology_of_Critical_Patient_with_Novel_Coronavirus_Pneumonia_COVID-19_Pulmonary_Fibrosis_and_Vascular_Changes_including_Microthrombosis_Formation
- See also: Generalized odds ratios for ordinal data — https://www.semanticscholar.org/paper/Generalized-Odds-Ratios-for-Ordinal-Data-Agresti/f7ac23e686de751706146f8dd926d1f03d1b0255

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated early and never unblinded. With only 2 subjects, statistical significance could never be demonstrated. Therefore, Arm/Group randomization information is not available.
Groups:
- All Study Participants: 1. TNKase (0.25 mg/kg) bolus as a sterile, lyophilized powder, diluted with 10mL sterile water, and administered as a 5-second bolus; AND standard of care anticoagulation therapy (enoxaparin or heparin).
     OR
  2. Placebo-to-match-TNKase bolus as a sterile, lyophilized powder, diluted with 10mL sterile water, and administered as a 5-second bolus; AND standard of care anticoagulation therapy (enoxaparin or heparin).
Period: Overall Study
Arm/Group | All Study Participants
Started | 2
Completed | 1
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The study was terminated early and never unblinded. With only 2 subjects, statistical significance could never be demonstrated. Therefore, Arm/Group randomization information is not available.
Arm/Group | All Study Participants
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Improvement in Shock Index (Defined as Heart Rate Divided by Systolic Blood Pressure) 6 Hours After the TNK/Placebo Bolus.
Description: For example, a patient may start with a heart rate of 100 beats/min and systolic blood pressure of 100 mm Hg (shock index = 1) and after therapy there may be an improvement where the heart rate is 90 beats/min, with systolic blood pressure of 110 mm Hg (shock index of 0.81), an improvement of 19%. A normal shock index is between 0.5 and 0.7 in healthy patients.
Time Frame: 6 hours post TNK/placebo infusion
Population: as for baseline characteristics
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: 1. Clinical Status at 24 Hours After Administration of TNK / Placebo Based Upon 7-point Scale.
Description: Assessment of patient status using an ordinal scale will be recorded at baseline and once daily in the morning while hospitalized.
  Level 1: Discharged (or "ready for discharge" on ambient air or < 2L suppl O2) Level 2: Non-ICU hospital ward (or "ready for hospital ward") not requiring suppl O2 Level 3: Non-ICU hospital ward (or "ready for hospital ward") requiring suppl O2 Level 4. ICU or non-ICU, requiring non-invasive ventilation or high-flow O2 Level 5. ICU, requiring intubation and mechanical ventilation Level 6: ICU, requiring ECMO or mechanical ventilation and additional organ support (e.g. vasopressors, renal replacement therapy) Level 7: Death
Time Frame: 24 +/- 6 hours post TNK/placebo infusion.
Population: as for baseline characteristics
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: The study not unblinded. All data was entered in treatment fields.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Attributable to COVID-19 Pneumonia
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) — Attributable to SOC anticoagulation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to enrollment being slower than anticipated, with study enrollment highly dependent upon COVID-19 surge patterns. We were otherwise hopeful to enroll and complete all assessments for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT04558125/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT04558125/ICF_001.pdf